CLINICAL TRIAL: NCT04357704
Title: Improved Speech Recognition Performance in Noise by Encoding Binaural Spatial Cues to the Cochlear Implant User.
Acronym: APPIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay in setting up the study.
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PIC_10
Record Dates: First submitted 2018-11-27; First posted 2020-04-22 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss, Cochlear
Keywords: Iteraural Time Difference
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral cochlear implant recipients (Experimental)
  Interventions: Other: S0N0; Other: S0N500; Other: S-500N500; Other: S0N1000; Other: S0Nuncorr
- normal hearing listners (Active Comparator)
  Interventions: Other: S0N0; Other: S0N500; Other: S-500N500; Other: S0N1000; Other: S0Nuncorr

INTERVENTIONS:
Other: S0N0 — (no ITD)
Other: S0N500 — (ITD +500µs on noise)
Other: S-500N500 — (ITD -500µs on signal and +500 µs on noise)
Other: S0N1000 — (ITD + 1000 µs on noise)
Other: S0Nuncorr — (no ITD cue, with uncorrelated stimulation frame)

SUMMARY:
The aim of the study is to evaluate the interaural time difference (ITD) benefit in patients with bilateral cochlear implants and to assess speech performance in noisy conditions compared to normal hearing listeners. Half of participants are bilateral cochlear implants users, while the other are normal hearing listeners.

DETAILED DESCRIPTION:
Listening in noisy environments is part of everyday life, it is based on binaural phenomena such as spatial localization.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in local language
* Normal hearing listener:
* pure tone threshold > 25dB from 125Hz to 12kHz
* Cochlear implant recipient
* bilaterally implanted 6 months at least, the second implant should be implanted 6 months at least before participant inclusion
* Digisonic SP® cochlear implants user

Exclusion Criteria:

* binaural sensitivity threshold < 1000µs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
speech reception threshold (SRT) in bilateral cochlear implant user with ITD cue | day 0
  SRT is used as an outcome measure to quantify the acuity for speech perception in noise with Interaural Time Difference between the two ears. Signal recognition in a background noise is assessed the following conditions S0N0, S0N500, S0N1000, S-500N500 et S0Nuncorr. The noise level is constant at 65 dB SPL, the signal level is modified in the adaptive procedure in order to converge towards a score of 50% of correct response.

SECONDARY OUTCOMES:
speech reception threshold (SRT) in bilateral cochlear implant user without ITD cue and in normal hearing listeners | day 0
  SRT is used as an outcome measure to quantify the acuity for speech perception in noise without Interaural Time Difference between the two ears.
ITD sensitivity in bilateral cochlear implant user | day 0
  Speech signal and noise are presented at 65dB SPL. Participant adjusts the Interaural Time Difference between the speech signal and noise between -1000 and +1000µs. Participant moves the cursor on the interface until he/she hears a difference in sound.
Preferred jitter in bilateral cochlear implant user | day 0
  Speech signal and noise are presented at 65dB SPL. Participant adjusts the jitter of the train pulse timing from 0 to +1000µs to improve the Interaural Time Difference.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guevara, MD, Principal Investigator — Hospital University Nice-IUFC; Alexis Bozorg-Grayeli, MD, Principal Investigator — Hospital University Dijon-François Mitterrand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: oticon medical website — http://www.oticonmedical.com